CLINICAL TRIAL: NCT00695825
Title: Postprandial Effects of a Low vs. a High Glycemic Index Food Product on Metabolic Risk Markers in Lean and Obese Subjects
Brief Title: Effects the Glycemic Index on Metabolic Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Ronald P. Mensink, Prof., Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 073101
Record Dates: First submitted 2008-06-04; First posted 2008-06-12 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Experimental): Consumption of low GI food product on day 1 Consumption of high GI food product on day 2
  Interventions: Dietary Supplement: Low GI+high GI
- A2 (Experimental): Consumption of high GI food product on day 1 Consumption of low GI food product on day 2
  Interventions: Dietary Supplement: High GI+low GI

INTERVENTIONS:
Dietary Supplement: Low GI+high GI — Consumption of low GI food product on day 1 Consumption of high GI food product on day 2
  Arms: A1
Dietary Supplement: High GI+low GI — Consumption of high GI food product on day 1 Consumption of low GI food product on day 2
  Arms: A2

SUMMARY:
Recent population studies have shown that the glycemic index (GI) of food products is positively associated with the risk of developing type 2 diabetes and cardiovascular disease (CVD). In the pathogenesis of type 2 diabetes and CVD, inflammatory processes play a pivotal role. In a previous intervention study (11 weeks), however, we found no effects of lower-GI vs. higher-GI diets on fasting inflammatory markers in subjects with increased risk of developing the metabolic syndrome. People, however, spent most of their time in the postprandial period. Therefore, there is a need to study the postprandial effects of low-GI vs. high-GI diets. In addition, it needs to be emphasized the GI is derived from studies in lean subjects, while especially overweight and obese people suffer from metabolic aberrations related to the development of type 2 diabetes and CVD. AIM: To investigate in obese subjects the postprandial effects of a low-GI vs. high-GI food product on metabolic risk markers. A second research objective is to compare these effects with those in lean subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy and obese men

Exclusion Criteria:

* smoking

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04-01 (Actual); Primary Completion 2006-11-30 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
inflammation markers | postprandial effect

SECONDARY OUTCOMES:
glucose response | postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Vrolix, PhD, Principal Investigator — Maastricht University
Locations (1):
- University Maastricht, Maastricht, Netherlands